CLINICAL TRIAL: NCT04949828
Title: Observational Study Assessing for Effect of CREON on Symptoms of Exocrine Pancreatic Insufficiency (EPI) in Patients With EPI Due to Chronic Pancreatitis (CP)
Brief Title: Effect of CREON on Exocrine Pancreatic Insufficiency (EPI) Symptoms
Acronym: CisCP
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-238
Record Dates: First submitted 2021-06-21; First posted 2021-07-02 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Chronic Pancreatitis
Keywords: Chronic pancreatitis; Exocrine Pancreatic Insufficiency; CREON; pancrelipase; ABT-SLV245
MeSH Terms: conditions — Pancreatitis, Chronic; Exocrine Pancreatic Insufficiency | interventions — Pancrelipase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants on CREON
  Interventions: Drug: CREON

INTERVENTIONS:
Drug: CREON — Oral Capsules
  Other Names: pancrelipase; ABT-SLV245

SUMMARY:
Exocrine Pancreatic Insufficiency (EPI) is a condition where pancreatic enzyme quantity or activity is reduced below threshold needed for normal digestion. Symptoms include bloating, flatulence, diarrhea and steatorrhea. This is an observational study assessing for effect of CREON on symptoms of EPI in participants with EPI due to chronic pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Medical history of chronic pancreatitis (CP).
* Diagnosis of Exocrine Pancreatic Insufficiency (EPI).

Exclusion Criteria:

--History of cystic fibrosis, pancreatic cancer, pancreatic surgery, gastric bypass surgery, extensive bowel surgery, inflammatory bowel disease, celiac disease, irritable bowel syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with medical diagnosis of chronic pancreatitis (CP) and exocrine pancreatic insufficiency (EPI)
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Change in Score of EPI Symptoms Domain Using an EPI Patient-Reported Outcomes Questionnaire | Up to 1 month

SECONDARY OUTCOMES:
Change in T-scores for Patient-Reported Outcomes Measurement and Information System(PROMIS) Questionnaires for Anxiety, Depression, and Fatigue | Up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (6):
- United States (6):
  - Stanford University School of Med /ID# 229530, Stanford, California
  - University of Florida - Archer /ID# 227057, Gainesville, Florida
  - John Hopkins University /ID# 227061, Baltimore, Maryland
  - NYU Langone Health /ID# 230818, New York, New York
  - The Ohio State University Wexner Medical Center /ID# 227844, Columbus, Ohio
  - Baylor College of Medicine - Baylor Medical Center /ID# 227067, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related info — https://www.rxabbvie.com/